CLINICAL TRIAL: NCT00959049
Title: A Phase III, Randomized, Observer-blind, Multi-center, Noninferiority Comparison of the Immune Response of CSL Limited's Influenza Virus Vaccine Compared to a US Licensed Trivalent Inactivated Split-Virion Influenza Vaccine in a Pediatric Population Aged Greater Than or Equal to 6 Months to Less Than 18 Years.
Brief Title: A Study to Determine the Immunogenicity and Safety Profile of CSL Limited's Influenza Virus Vaccine Compared to a US Licensed Comparator Influenza Virus Vaccine in a Pediatric Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CSLCT-USF-07-36
Record Dates: First submitted 2009-08-12; First posted 2009-08-14 (Estimated); Results first posted 2011-07-29 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Afluria; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Afluria Cohort A (Experimental): Age 6 months to < 3 years
  Interventions: Biological: CSL's Influenza Virus Vaccine (Afluria)
- Afluria Cohort B (Experimental): Age 3 to < 9 years
  Interventions: Biological: CSL's Influenza Virus Vaccine (Afluria)
- Afluria Cohort C (Experimental): Age 9 to < 18 years
  Interventions: Biological: CSL's Influenza Virus Vaccine (Afluria)
- Fluzone Cohort A (Active Comparator): Age 6 months to < 3 years
  Interventions: Biological: Influenza Virus Vaccine (Fluzone)
- Fluzone Cohort B (Active Comparator): Age 3 to < 9 years
  Interventions: Biological: Influenza Virus Vaccine (Fluzone)
- Fluzone Cohort C (Active Comparator): Age 9 to < 18 years
  Interventions: Biological: Influenza Virus Vaccine (Fluzone)

INTERVENTIONS:
Biological: CSL's Influenza Virus Vaccine (Afluria) — 0.25 mL (one or two doses) or 0.5 mL (one or two doses) by intramuscular injection as directed by immunization guidelines
  Arms: Afluria Cohort A; Afluria Cohort B; Afluria Cohort C
Biological: Influenza Virus Vaccine (Fluzone) — 0.25 mL (one or two doses) or 0.5 mL (one or two doses) by intramuscular injection as directed by immunization guidelines
  Arms: Fluzone Cohort A; Fluzone Cohort B; Fluzone Cohort C

SUMMARY:
The purpose of this study is to determine the immunogenicity and safety profile of CSL Limited's Influenza Virus Vaccine compared to a US licensed comparator Influenza Virus Vaccine in a pediatric population aged greater than or equal to 6 months to less than 18 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female participants aged ≥ 6 calendar months to < 18 years at the time of the first study vaccination.
* For participants aged ≥ 6 months to < 9 years, born after a normal gestation period (between 36 and 42 weeks).
* Females of childbearing potential (i.e., ovulating, pre-menopausal, not surgically sterile) must be abstinent or be willing to use a medically accepted contraceptive regimen for at least 2 months after vaccination. Females aged ≥ 9 years must also return a negative urine pregnancy test at enrollment.

Exclusion Criteria:

* Known hypersensitivity to a previous dose of influenza vaccine or allergy to eggs, chicken protein, neomycin, polymyxin, or any components of the Study Vaccine.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1474 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director Vaccines, Study Director — Seqirus
Locations (21):
- United States (21):
  - Chandler, Arizona
  - Harrisburg, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Mountain Home, Arkansas
  - Melbourne, Florida
  - Bardstown, Kentucky
  - Omaha, Nebraska
  - Binghamton, New York
  - Elmira, New York
  - Cincinnati Children's Hospital Medical Center- Division of Infectious Disease, Cincinnati, Ohio
  - Warr Acres, Oklahoma
  - UPMC / Community Medicine Inc, Greenville, Pennsylvania
  - Pediatric Associates of Latrobe, Latrobe, Pennsylvania
  - Pediatric Alliance Greentree Division, Pittsburgh, Pennsylvania
  - South Hills Pediatrics, Pittsburgh, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Salt Lake City, Utah
  - South Jordan, Utah
  - Burke, Virginia
  - Vienna, Virginia

REFERENCES:
- [Derived] Brady RC, Hu W, Houchin VG, Eder FS, Jackson KC, Hartel GF, Sawlwin DC, Albano FR, Greenberg M. Randomized trial to compare the safety and immunogenicity of CSL Limited's 2009 trivalent inactivated influenza vaccine to an established vaccine in United States children. Vaccine. 2014 Dec 12;32(52):7141-7. doi: 10.1016/j.vaccine.2014.10.024. Epub 2014 Oct 29. PMID 25454878

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled into this study during the autumn of 2009 at 23 sites in the US.
Pre-assignment Details: A total of 1474 participants were enrolled, vaccinated and analyzed.
Groups:
- Afluria Cohort A: Age 6 months to < 3 years. Participants received one of two doses of the 2009/2010 influenza season formulation of Afluria.
- Afluria Cohort B: Age 3 to < 9 years. Participants received one or two doses of the 2009/2010 influenza season formulation of Afluria.
- Afluria Cohort C: Age 9 to < 18 years. Participants received one or two doses of the 2009/2010 influenza season formulation of Afluria.
- Fluzone Cohort A: Age 6 months to < 3 years. Participants received one of two doses of the 2009/2010 influenza season formulation of Fluzone.
- Fluzone Cohort B: Age 3 to < 9 years. Participants received one of two doses of the 2009/2010 influenza season formulation of Fluzone.
- Fluzone Cohort C: Age 9 to < 18 years. Participants received one of two doses of the 2009/2010 influenza season formulation of Fluzone.
Period: Overall Study
Arm/Group | Afluria Cohort A | Afluria Cohort B | Afluria Cohort C | Fluzone Cohort A | Fluzone Cohort B | Fluzone Cohort C
Started | 231 | 254 | 254 | 228 | 257 | 250
Completed | 213 | 247 | 253 | 217 | 248 | 249
Not Completed | 18 | 7 | 1 | 11 | 9 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 17 | 5 | 1 | 10 | 9 | 1
Not completed — Contraindicated medication | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Afluria Cohort A | Afluria Cohort B | Afluria Cohort C | Fluzone Cohort A | Fluzone Cohort B | Fluzone Cohort C | Total
Number analyzed (Participants) | 231 | 254 | 254 | 228 | 257 | 250 | 1474
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 231 | 254 | 254 | 228 | 257 | 250 | 1474
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.94 (0.667) | 5.93 (1.725) | 12.98 (2.388) | 1.96 (0.673) | 5.82 (1.748) | 12.86 (2.474) | 7.06 (4.855)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 140 | 121 | 101 | 127 | 120 | 728
  Male | 112 | 114 | 133 | 127 | 130 | 130 | 746
Region of Enrollment [Number; unit: participants]
  United States | 231 | 254 | 254 | 228 | 257 | 250 | 1474

OUTCOME MEASURES:

1. Secondary Outcome: Frequency and Intensity of Local and Systemic Solicited Symptoms, Cohort A (6 Months to < 3 Years)
Time Frame: 7 days after each vaccination
Population: Safety population; Afluria Cohort A receiving 2 doses N=96, Fluzone Cohort A receiving 2 doses N=110
Measure: Number; unit: Participants
Arm/Group | Afluria Cohort A | Fluzone Cohort A
Number analyzed (Participants) | 229 | 228
Participants
  Any local solicited symptom post-dose 1 | 116 | 100
  Any pain (post dose 1) | 98 | 78
  Grade 3 pain (post dose 1) | 1 | 0
  Any redness (> 0 mm) (post dose 1) | 53 | 53
  Grade 3 redness (> 30 mm) (post dose 1) | 0 | 1
  Any swelling (> 0 mm) (post dose 1) | 30 | 26
  Grade 3 swelling (> 30 mm) (post dose 1) | 1 | 0
  Any local solicited symptom post-dose 2 | 30 | 32
  Any pain (post dose 2) | 28 | 22
  Grade 3 pain (post dose 2) | 0 | 0
  Any redness (> 0 mm) (post dose 2) | 15 | 22
  Grade 3 redness (> 30 mm) (post dose 2) | 1 | 0
  Any swelling (> 0 mm) (post dose 2) | 9 | 7
  Grade 3 swelling (> 30 mm) (post dose 2) | 0 | 0
  Any systemic solicited symptom, post dose 1 | 171 | 121
  Any fever ≥ 99.5°F ax or≥ 100.4°F oral, dose1 | 85 | 31
  Grade 3 fever > 103.1°F ax or> 104.0°F oral, dose1 | 6 | 0
  Any nausea/vomiting, dose 1 | 27 | 17
  Grade 3 nausea/vomiting prevented activities,dose1 | 22 | 6
  Any diarrhea, dose 1 | 61 | 54
  Grade 3 diarrhea prevented activities, dose 1 | 4 | 3
  Any loss of appetite, dose 1 | 73 | 45
  Grade3 loss of appetite prevented activities dose1 | 3 | 1
  Any irritability, dose 1 | 134 | 85
  Grade 3 irritability prevented activities dose 1 | 10 | 5
  Any systemic solicited symptom post-dose 2 | 48 | 44
  Any fever ≥ 99.5°F ax or≥ 100.4°F oral, dose 2 | 14 | 15
  Grade 3 fever > 103.1°F ax or> 104.0°F oral, dose2 | 1 | 0
  Any nausea/vomiting, dose 2 | 4 | 8
  Grade3 nausea/vomiting prevented activities, dose2 | 2 | 0
  Any diarrhea, dose 2 | 17 | 16
  Grade3 diarrhea (prevented activities), dose 2 | 1 | 0
  Any loss of appetite, dose 2 | 15 | 14
  Grade3 loss of appetite prevented activities dose2 | 1 | 0
  Any irritability, dose 2 | 38 | 31
  Grade 3 irritability prevented activities, dose 2 | 1 | 0

2. Secondary Outcome: Frequency and Intensity of Local and Systemic Solicited Symptoms, Cohort B
Time Frame: 7 days after each vaccination
Population: Safety population; Afluria cohort B receiving 2 doses N=68, Fluzone cohort B receiving 2 doses N=78
Measure: Number; unit: Participants
Arm/Group | Afluria Cohort B | Fluzone Cohort B
Number analyzed (Participants) | 252 | 255
Participants
  Any local solicited symptom post-dose 1 | 164 | 152
  Any pain, post dose 1 | 149 | 131
  Grade 3 pain, post dose 1 | 1 | 4
  Any redness (> 0 mm), post dose 1 | 59 | 60
  Grade 3 redness (> 30 mm), post dose 1 | 7 | 4
  Any swelling (> 0 mm), post dose 1 | 36 | 43
  Grade 3 swelling (> 30 mm), post dose 1 | 6 | 2
  Any local solicited symptom post-dose 2 | 24 | 26
  Any pain, post dose 2 | 23 | 23
  Grade 3 pain, post dose 2 | 0 | 0
  Any redness (> 0 mm), post dose 2 | 5 | 13
  Grade 3 redness (> 30 mm), post dose 2 | 0 | 0
  Any swelling (> 0 mm), post dose 2 | 4 | 11
  Grade 3 swelling (> 30 mm), post dose 2 | 0 | 0
  Any systemic solicited symptom post-dose 1 | 140 | 113
  Any fever ≥ 99.5°F ax or ≥ 100.4°F oral, dose 1 | 55 | 24
  Grade 3 fever > 103.1°F ax or > 104.0°F oral dose1 | 3 | 1
  Any nausea/vomiting, dose 1 | 33 | 20
  Grade3 nausea/vomiting prevented activities, dose1 | 2 | 1
  Any diarrhea, dose 1 | 17 | 24
  Grade 3 diarrhea (prevented activities), dose 1 | 0 | 0
  Any malaise, dose 1 | 72 | 34
  Grade 3 malaise (prevented activities), dose 1 | 9 | 1
  Any headache, dose 1 | 54 | 41
  Grade 3 headache (prevented activities), dose 1 | 5 | 0
  Any myalgia, dose 1 | 82 | 63
  Grade 3 myalgia (prevented activities), dose 1 | 1 | 1
  Any systemic solicited symptom post-dose 2 | 17 | 18
  Any fever ≥ 99.5°F ax or ≥ 100.4°F oral dose 2 | 4 | 5
  Grade3 fever > 103.1°F ax or> 104.0°F oral, dose 2 | 1 | 0
  Any nausea/vomiting, dose 2 | 2 | 4
  Grade3 nausea/vomiting prevented activities ,dose2 | 1 | 0
  Any diarrhea, dose 2 | 6 | 5
  Grade 3 diarrhea (prevented activities), dose 2 | 0 | 0
  Any malaise, dose 2 | 6 | 6
  Grade 3 malaise (prevented activities), dose 2 | 0 | 0
  Any headache, dose 2 | 6 | 8
  Grade 3 headache (prevented activities), dose 2 | 0 | 0
  Any myalgia, dose 2 | 7 | 12
  Grade 3 myalgia (prevented activities), dose 2 | 0 | 0

3. Secondary Outcome: Frequency and Intensity of Local and Systemic Solicited Symptoms, Cohort C
Time Frame: 7 days after vaccination
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Afluria Cohort C | Fluzone Cohort C
Number analyzed (Participants) | 254 | 250
Participants
  Any local solicited symptom post-dose 1 | 174 | 169
  Any pain | 167 | 151
  Grade 3 pain (prevented activities) | 1 | 4
  Any redness (> 0 mm) | 43 | 43
  Grade 3 redness (> 30 mm) | 1 | 3
  Any swelling (> 0 mm) | 39 | 41
  Grade 3 swelling (> 30 mm) | 4 | 7
  Any systemic solicited symptom post-dose 1 | 144 | 126
  Any fever (≥ 99.5°F ax or ≥ 100.4°F oral) | 16 | 10
  Grade 3 fever (> 103.1°F ax or > 104.0°F oral) | 2 | 0
  Any nausea/vomiting | 23 | 24
  Grade 3 nausea/vomiting (prevented activities) | 3 | 3
  Any diarrhea | 20 | 25
  Grade 3 diarrhea (prevented activities) | 1 | 0
  Any malaise | 55 | 51
  Grade 3 malaise (prevented activities) | 10 | 3
  Any headache | 69 | 66
  Grade 3 headache (prevented activities) | 7 | 3
  Any myalgia | 101 | 93
  Grade 3 myalgia (prevented activities) | 5 | 4

4. Primary Outcome: Geometric Mean Titer 30 Days After the Last Study Vaccination
Time Frame: 30 days after the last study vaccination
Population: Per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Afluria Cohort A | Afluria Cohort B | Afluria Cohort C | Fluzone Cohort A | Fluzone Cohort B | Fluzone Cohort C
Number analyzed (Participants) | 195 | 229 | 230 | 201 | 236 | 233
Titers
  H1N1 (A/Brisbane/59/2007) | 235.44 [199.67 to 277.61] | 345.50 [295.54 to 403.92] | 652.99 [566.91 to 752.14] | 227.19 [188.39 to 273.98] | 351.88 [303.29 to 408.25] | 652.17 [569.59 to 746.73]
  H3N2 ( A/Uruguay/716/2007) | 309.19 [253.49 to 377.13] | 909.22 [772.67 to 1069.90] | 948.86 [824.88 to 1091.46] | 340.49 [283.98 to 408.25] | 870.34 [751.62 to 1007.80] | 1069.7 [934.77 to 1224.11]
  B (B/Brisbane/60/2008) | 73.46 [59.32 to 90.97] | 122.71 [102.55 to 146.83] | 107.92 [71.77 to 126.91] | 57.92 [46.92 to 71.49] | 104.91 [88.67 to 123.42] | 126.99 [107.53 to 149.97]

5. Primary Outcome: Percentage of Participants With Seroconversion 30 Days After the Last Study Vaccination
Description: Seroconversion rate was defined as the proportion of participants with either a titer of less than 1:10 before vaccination achieving a HI antibody titer of 1:40 or more after vaccination, or a HI titer of 1:10 or more before vaccination achieving a four-fold or greater increase in HI titer after vaccination.
Time Frame: 30 days after the last study vaccination
Population: Per-Protocol Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afluria Cohort A | Afluria Cohort B | Afluria Cohort C | Fluzone Cohort A | Fluzone Cohort B | Fluzone Cohort C
Number analyzed (Participants) | 195 | 229 | 230 | 201 | 236 | 233
Percentage of participants
  H1N1 (A/Brisbane/59/2007) | 84 [78 to 89] | 66 [59 to 72] | 64 [57 to 70] | 74 [67 to 80] | 64 [58 to 70] | 61 [55 to 68]
  H3N2 ( A/Uruguay/716/2007) | 83 [77 to 88] | 71 [65 to 77] | 72 [66 to 78] | 85 [79 to 90] | 74 [68 to 80] | 73 [66 to 78]
  B (B/Brisbane/60/2008) | 67 [60 to 73] | 73 [67 to 79] | 67 [31 to 73] | 61 [54 to 68] | 76 [70 to 82] | 73 [67 to 79]

6. Secondary Outcome: Frequency and Intensity of Unsolicited Adverse Events (UAEs)
Description: UAE stands for Unsolicited Adverse Events
Time Frame: 30 days after each vaccination
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Afluria Cohort A | Afluria Cohort B | Afluria Cohort C | Fluzone Cohort A | Fluzone Cohort B | Fluzone Cohort C
Number analyzed (Participants) | 229 | 252 | 254 | 228 | 255 | 250
Participants
  Any | 123 | 100 | 88 | 112 | 84 | 70
  Grade 3 | 28 | 25 | 17 | 24 | 22 | 16
  Any related | 37 | 24 | 20 | 16 | 18 | 14

7. Secondary Outcome: New Onset of Chronic Illnesses (NOCIs)
Description: New onset of chronic illness after any vaccine dose. A new onset of chronic illness was defined as the diagnosis of a new medical condition which was chronic in nature, including those potentially controllable by medication (e.g., diabetes, asthma).
Time Frame: 6 months after last study vaccination
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Afluria Cohort A | Afluria Cohort B | Afluria Cohort C | Fluzone Cohort A | Fluzone Cohort B | Fluzone Cohort C
Number analyzed (Participants) | 229 | 252 | 254 | 228 | 255 | 250
Participants
  Total number of participants with NOCI | 2 | 0 | 2 | 2 | 1 | 0
  Number of participants with related NOCI | 0 | 0 | 0 | 0 | 0 | 0
  Asthma | 1 | 0 | 2 | 1 | 0 | 0
  Von Willebrand's Disease | 1 | 0 | 0 | 0 | 0 | 0
  Eczema | 0 | 0 | 0 | 1 | 0 | 0
  Attention deficit disorder | 0 | 0 | 0 | 0 | 1 | 0

8. Secondary Outcome: Serious Adverse Events (SAEs)
Time Frame: 6 months after last study vaccination
Population: Safety Population
Measure: Number; unit: Participants
Groups:
- Fluzone Cohort C: Age 3 to < 9 years
Arm/Group | Afluria Cohort A | Afluria Cohort B | Afluria Cohort C | Fluzone Cohort A | Fluzone Cohort B | Fluzone Cohort C
Number analyzed (Participants) | 229 | 252 | 254 | 228 | 255 | 250
Participants
  Number of participants with SAEs | 4 | 2 | 2 | 4 | 0 | 0
  Number of participants with related SAEs | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Duration of Local and Systemic Solicited Symptoms, Cohort A (6 Months to < 3 Years)
Time Frame: 7 days after each vaccination
Population: Safety population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Afluria Cohort A | Fluzone Cohort A
Number analyzed (Participants) | 229 | 228
Days
  Any pain post-dose 1 | 1.57 (0.952) | 1.43 (0.728)
  Any redness (> 0 mm), post dose 1 | 2.09 (1.405) | 2.22 (1.939)
  Any swelling (> 0 mm), post dose 1 | 3.13 (2.930) | 2.00 (1.569)
  Any pain post-dose 2 | 1.54 (0.793) | 1.45 (0.739)
  Any redness (> 0 mm), post dose 2 | 1.80 (1.014) | 1.73 (0.935)
  Any swelling (> 0 mm), post dose 2 | 1.67 (0.707) | 1.57 (0.787)
  Any fever dose 1 (≥ 99.5°F ax or ≥ 100.4°F oral) | 1.38 (0.869) | 1.49 (0.989)
  Any nausea/vomiting, post dose 1 | 1.42 (1.119) | 1.29 (1.042)
  Any diarrhea, post dose 1 | 2.23 (2.157) | 2.16 (2.189)
  Any loss of appetite, post dose 1 | 2.61 (3.695) | 2.85 (4.458)
  Any irritability, post dose 1 | 2.26 (2.858) | 2.64 (3.825)
  Any fever dose 2 (≥ 99.5°F ax or ≥ 100.4°F oral) | 1.80 (1.146) | 1.81 (1.559)
  Any nausea/vomiting, post dose 2 | 2.50 (1.291) | 1.78 (1.093)
  Any diarrhea, post dose 2 | 2.83 (2.431) | 2.44 (2.332)
  Any loss of appetite, post dose 2 | 2.47 (1.586) | 2.33 (1.447)
  Any irritability, post dose 2 | 2.31 (1.732) | 2.17 (1.543)

10. Secondary Outcome: Duration of Local and Systemic Solicited Symptoms, Cohort B
Time Frame: 7 days after each vaccination
Population: Safety population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Afluria Cohort B | Fluzone Cohort B
Number analyzed (Participants) | 252 | 255
Days
  Any pain post-dose 1 | 1.89 (1.138) | 1.89 (1.337)
  Any redness (> 0 mm), post dose 1 | 2.32 (1.621) | 2.10 (2.014)
  Any swelling (> 0 mm), post dose 1 | 2.39 (2.021) | 2.09 (1.273)
  Any pain post-dose 2 | 1.96 (1.637) | 1.65 (0.775)
  Any redness (> 0 mm), post dose 2 | 2.40 (2.191) | 1.77 (1.235)
  Any swelling (> 0 mm), post dose 2 | 3.00 (2.160) | 1.69 (1.251)
  Any fever dose 1 (≥ 99.5°F ax or ≥ 100.4°F oral) | 1.45 (1.032) | 1.40 (0.707)
  Any nausea/vomiting, post dose 1 | 1.27 (0.719) | 1.43 (1.165)
  Any diarrhea, post dose 1 | 2.89 (4.988) | 1.44 (1.044)
  Any malaise, post dose 1 | 1.86 (1.324) | 1.74 (1.094)
  Any headache, post dose 1 | 1.50 (0.770) | 1.66 (1.328)
  Any myalgia, post dose 1 | 1.72 (1.007) | 1.63 (1.009)
  Any fever dose 2 (≥ 99.5°F ax or ≥ 100.4°F oral) | 1.50 (0.577) | 1.00 (0.000)
  Any nausea/vomiting, post dose 2 | 1.00 (0.000) | 1.20 (0.447)
  Any diarrhea, post dose 2 | 1.33 (0.816) | 2.20 (0.447)
  Any malaise, post dose 2 | 1.83 (1.602) | 1.71 (0.756)
  Any headache, post dose 2 | 1.00 (0.000) | 1.30 (0.483)
  Any myalgia, post dose 2 | 2.00 (1.528) | 1.54 (0.660)

11. Secondary Outcome: Duration of Local and Systemic Solicited Symptoms, Cohort C
Time Frame: 7 days after vaccination
Population: Safety population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Afluria Cohort C | Fluzone Cohort C
Number analyzed (Participants) | 254 | 250
Days
  Any pain | 1.96 (1.087) | 1.99 (1.136)
  Any redness (> 0 mm) | 2.02 (1.669) | 2.38 (1.992)
  Any swelling (> 0 mm) | 1.75 (1.171) | 2.38 (1.724)
  Any fever (≥ 99.5°F ax or ≥ 100.4°F oral) | 1.82 (1.590) | 3.10 (2.644)
  Any nausea/vomiting | 1.36 (0.569) | 2.88 (3.791)
  Any diarrhea | 1.18 (0.395) | 1.36 (0.911)
  Any malaise | 2.09 (1.487) | 2.82 (3.449)
  Any headache | 1.77 (1.443) | 2.05 (1.945)
  Any myalgia | 1.76 (1.100) | 2.11 (1.491)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 180 days after the last study vaccination.
Arm/Group | Afluria Cohort A | Afluria Cohort B | Afluria Cohort C | Fluzone Cohort A | Fluzone Cohort B | Fluzone Cohort C
Serious Adverse Events (participants affected / at risk) | 4/229 | 3/252 | 2/254 | 4/228 | 0/255 | 0/250
Other Adverse Events (participants affected / at risk) | 210/231 | 216/254 | 214/254 | 187/228 | 202/257 | 202/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Afluria Cohort A (N=229) | Afluria Cohort B (N=252) | Afluria Cohort C (N=254) | Fluzone Cohort A (N=228) | Fluzone Cohort B (N=255) | Fluzone Cohort C (N=250)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncitial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Afluria Cohort A (N=231) | Afluria Cohort B (N=254) | Afluria Cohort C (N=254) | Fluzone Cohort A (N=228) | Fluzone Cohort B (N=257) | Fluzone Cohort C (N=250)
Pain at the injection site (General disorders) | 107/229 | 157/252 | 167 | 89 | 134/255 | 151
Redness at the injection site (General disorders) | 60/229 | 62/252 | 43 | 60 | 67/255 | 43
Swelling at the injection site (General disorders) | 34/229 | 38/252 | 39 | 29 | 50/255 | 41
Fever (General disorders) | 91/229 | 58/252 | 16 | 42 | 29/255 | 10
Nausea/vomiting (Gastrointestinal disorders) | 31/229 | 35/252 | 23 | 23 | 24/255 | 24
Diarrhea (Gastrointestinal disorders) | 69/229 | 22/252 | 20 | 63 | 27/255 | 25
Loss of appetite (General disorders) | 79/229 | 0/252 | 0 | 54 | 0/255 | 0
Irritability (General disorders) | 142/229 | 0/252 | 0 | 99 | 0/255 | 0
Malaise (General disorders) | 0/229 | 74/252 | 55 | 0 | 37/255 | 51
Headache (General disorders) | 0/229 | 58/252 | 69 | 0 | 45/255 | 66
Myalgia (General disorders) | 0/229 | 87/252 | 101 | 0 | 66/255 | 93
Upper respiratory tract infection (Infections and infestations) | 9/229 | 6/252 | 4 | 14 | 5/255 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 39/229 | 40/252 | 19 | 31 | 33/255 | 17
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 25/229 | 14/252 | 5 | 24 | 10/255 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 14/229 | 8/252 | 16 | 11 | 4/255 | 6
Diarrhea (Gastrointestinal disorders) | 10/229 | 3/252 | 4 | 13 | 3/255 | 1
Pyrexia (General disorders) | 32/229 | 24/252 | 12 | 22 | 17/255 | 7
Headache (Nervous system disorders) | 6/229 | 6/252 | 17 | 3 | 8/255 | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4/229 | 7/252 | 19 | 2 | 6/255 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less